CLINICAL TRIAL: NCT05537337
Title: Multiphase Optimal Strategy To Improve Diet Quality-MOSTDQ (Aim 2)
Brief Title: Understanding Food Choices (Aim 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Eric A. Finkelstein, Professor, Duke-NUS Graduate Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: MOH-000263 (Aim 2)
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Diet Quality
Keywords: Multicomponent Intervention; Multiphase Optimization Strategy; Food Labels; Food Repositioning; Within-group Substitutes; Randomized Control Trial (RCT)

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Control Arm) (No Intervention): Participants will experience an unmodified version of NUSMart that is designed to replicate the traditional shopping experience of any online grocery shopping platform with details such as item description, brand, price, image, nutritional information etc.
- Arm 2 (Multicomponent Intervention Arm) (Experimental): Participants will experience a modified version of NUSMart with the multicomponent intervention enabled. This intervention consists of a subset of the combined interventions tested in Aim 1 namely, 1. Food labels (with the summary of healthiness of shopping baskets & targets), 2. Ordering and 3. Within Group Healthier Substitution.
  Interventions: Behavioral: Multicomponent Intervention

INTERVENTIONS:
Behavioral: Multicomponent Intervention — The multicomponent intervention consists of the following components (already described in the detailed description section):
  1. Food labels (with the summary of healthiness of shopping baskets & targets)
  2. Ordering
  3. Within Group Healthier Substitution
  Arms: Arm 2 (Multicomponent Intervention Arm)

SUMMARY:
This study aims to use the Multiphase Optimization Strategy (MOST) to build and optimize a multicomponent intervention that improves diet quality. The investigators have evaluated the effects of evidence-based public health interventions on consumers' diet quality via a web-based grocery store "NUSMart" as part of Aim 1 of this study. Considering that the goal is to identify promising interventions that may optimize online grocery platforms, the investigators used Aim 1's results to assemble a multicomponent intervention that would significantly affect diet quality: a combination of three behavioral nudges that include food labels & real-time feedback, ordering, and healthier substitute offers (a subset of the interventions examined in Aim 1). Aim 2 study aims to rigorously evaluate this multicomponent intervention.

DETAILED DESCRIPTION:
The important role that diet plays in health and disease is well established. Excessive intake of energy, saturated fat and sodium increase the risk of heart disease, diabetes and certain cancers. As a result, interventions aimed at encouraging healthier food consumption have been pursued by many countries. These can be broadly grouped into the following categories: price manipulations, food labelling, and behavioral nudges.

No study has previously assessed the potentially interactive effects of a multicomponent intervention that incorporates the strongest features of each intervention component while discarding those that do not meaningfully contribute to healthier consumption. That is the goal of this effort.

At part of the first stage of the MOST framework (Aim 1), the investigators evaluated the effects of evidence-based public health interventions on consumers' diet quality on a web-based grocery store "NUSMart". The investigators focused on the following four interventions: 1. Explicit Tax, 2. Food labels (with the summary of healthiness of shopping baskets & targets), 3. Ordering and 4. Within Group Healthier Substitution. Based on the study results, the investigators assembled a multicomponent intervention that consists of a subset of the above four interventions that may optimize online grocery platforms in terms of diet improvement.

The multicomponent intervention consists of the following components:

1. Food labels (with the summary of healthiness of shopping baskets & targets)- Food labels, called Nutri-Traffic-Lights (NTL), indicating whether food and beverage products were healthy, unhealthy or somewhere in between were designed for all products on NUSMart based on the Nutri-Score Nutrition Scoring System. These were supplemented with a video explaining the labels and a dynamic pie chart indicating the overall nutritional quality of the shopper's basket (updated in real time) known as MyCart summary.
2. Ordering- Healthier products, in terms of Nutri-Score Points, were displayed first within each category and subcategory.
3. Within Group Healthier Substitution- At checkout, up to 4 healthier substitutes were suggested for products in the shopper's cart based on the Nutri-Score Points of these products. Substitutes were from the same category as the product that was added to cart and were close to the original product in terms of price as well.

In this study (Aim 2), using a 2-arm randomized controlled trial, the investigators will test whether the assembled multicomponent intervention has a sustained positive effect on diet quality over 3 purchases over a 3-5-week period, wherein the purchased foods are delivered to the participants' homes.

Over the course of the study, participants will log into the NUSMart website once a week and will be asked to purchase their weekly groceries with a minimum spend of $59. Each participant will therefore shop a total of 3 times using the same version of NUSMart randomly assigned to them, during the study.

The investigators' hypotheses about the effects of the multicomponent intervention on diet quality, measured by the weighted (by the number of servings) average Nutri-Score Points (primary) of finalized shopping baskets, are as follows:

1. The multicomponent intervention will significantly improve diet quality as measured by the weighted Nutri-Score Points (primary), calories, sodium, sugar, and saturated fat per serving, which will be calculated based on all purchased products' total nutritional value.
2. The improvements in diet quality will be sustained through repeated shops where food is actually delivered, thus making it more likely that results are externally valid.

ELIGIBILITY:
Inclusion Criteria:

* Singapore resident
* Age 21 and above
* Must be the primary weekly grocery shopper in their household

Exclusion Criteria:

* Non-Singapore resident
* Less than 21 years old
* Non-primary grocery shopper in their household

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 487 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Diet Quality | After completion of data collection, an average of about 14 months
  Diet quality measured by the weighted (by the number of servings) average of all purchased products' Nutri-Score Points for the shopping trip. Nutri-Score Points is an individual dietary index based on the British Food Standard Agency Nutrient Profiling System. Nutri-Score points are calculated by scoring food and beverage products on a scale from -15 (healthiest) to 40 (least healthy) by subtracting the sum of Nutri-Score sub-points for healthier components (e.g., fiber, protein, percentage of fruits & vegetables) from the sum of Nutri-Score sub-points for less healthy components (e.g., energy, sugar, sodium, saturated fat). The final non-numeric grade, A to E, is determined based on carefully designed thresholds for these resulting Nutri-Score Points.

SECONDARY OUTCOMES:
Nutrients per serving | After completion of data collection, an average of about 14 months
  Average calories, sodium, sugar, and saturated fat per serving, which will be calculated based on all purchased products' total nutritional value.
Proportion of products for each Nutri-Traffic-Light (NTL) classification | After completion of data collection, an average of about 14 months
  The proportion of products eligible for each of the 3 classifications of the NTL (i.e., the green circle, the amber circle and the red stop-sign) respectively, of the purchased products.

OTHER OUTCOMES:
Mediators, Moderators and Covariates | After completion of data collection, an average of about 14 months
  We will run models both with and without including covariates that include demographic variables (e.g., age, minority status, income, BMI, sex, and household size) and measurements of health-status. To test the moderating effects of health-status, and education level, we will include interaction terms between the intervention arm and these variables.

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Finkelstein, PhD MHA, Principal Investigator — Duke-NUS Graduate Medical School
Locations (1):
- Duke-NUS Graduate Medical School, Singapore, Singapore

REFERENCES:
- [Derived] Shin S, Xiaoxi Y, Chakraborty B, Finkelstein EA. A Randomized Trial Using an Online Grocery Store to Evaluate a Multicomponent Digital Intervention to Improve Diet Quality. Am J Prev Med. 2025 Jul;69(1):107622. doi: 10.1016/j.amepre.2025.03.002. Epub 2025 Mar 20. PMID 40120994